CLINICAL TRIAL: NCT03938792
Title: An Open-Label Study in Adolescent and Adult Severe (Coagulation Factor Activity <1%) Hemophilia A Participants With or Without Inhibitors or Moderately Severe to Severe Hemophilia B Participants (Coagulation Factor Activity ≤2%) With or Without Inhibitors Comparing Standard Treatment to PF-06741086 Prophylaxis
Brief Title: Study of the Efficacy and Safety PF-06741086 in Adult and Teenage Participants With Severe Hemophilia A or Moderately Severe to Severe Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B7841005; 2018-003660-31 (EudraCT Number)
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Factor VIII; Factor IX; Inhibitors; Anti-Tissue Factor Pathway Inhibitor (TFPI); Subcutaneous (sc); Prophylaxis; On-Demand; BASIS; Inhibitor; SC; Subcutaneous; Injection; On demand; aTFPI; Anti-TFPI; Severe hemophilia; Severe bleeding; Hemophilia; PF-06741086; PF 06741086; Marstacimab
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Hemorrhage | interventions — marstacimab

STUDY DESIGN:
Intervention Model Description: This is a one way Cross-Over Prevention study with 1 Arm that has No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06741086 (Experimental): Participants will be assigned to treatment with PF-06741086 after a 6 month Observation Phase on their current hemophilia regimen.
  Interventions: Drug: PF-06741086

INTERVENTIONS:
Drug: PF-06741086 — 300 milligrams(mg) subcutaneous (sc) loading dose followed by 150 mg sq once weekly (qw). 300 mg sc qw is prescribed for participants who meet dose escalation criteria.

SUMMARY:
Treatment with PF-06741086 is anticipated to demonstrate a clinically relevant advantage and/or a major contribution to patient care in comparison to current methods of treatment for hemophilia A or B because it works differently than factor replacement products and will work in the presence of inhibitors. The potential for once weekly (QW) subcutaneous (SC) administration provides for treatment options in the absence of reliable vascular access, increased convenience and may enable better compliance. Combined, these qualities should result in a reduction of bleeding episodes.

ELIGIBILITY:
Inclusion Criteria

* Participants with a diagnosis of severe hemophilia A or moderately severe to severe hemophilia B with a minimum weight of 35 kg at screening.
* Participant or legally authorized representative, or participant's caregiver capable of giving signed informed consent (or minor assent, when applicable).

Participants who are enrolled into the Non-Inhibitor Cohort must also meet the following criteria:

* No detectable or documented history of inhibitors
* Participants on FVIII/FIX routine prophylaxis who have demonstrated at least 80% compliance with scheduled prophylaxis regimen during 6 months prior to enrollment and are willing to continue to receive routine prophylaxis treatment with FVIII/FIX replacement during the Observational Phase.
* Participants with on-demand treatment regimen with ≥6 acute bleeding episodes (spontaneous or traumatic) that required coagulation factor infusion during the 6 months period prior to enrollment and willing to continue to receive on demand treatment during the Observational Phase.

Participants who are enrolled into the Inhibitor Cohort must also meet the following criteria:

* Documentation of current high titer inhibitor (≥5 BU/mL) or current low titer inhibitor (<5 BU/mL) refractory to FVIII or FIX replacement and with FVIII or FIX recovery <60% of expected within previous 6 months prior to enrolment into the Observational Phase
* Hemophilia A participants with on-demand treatment regimen with ≥6 bleeding episodes or hemophilia B participants with ≥4 bleeding episodes (spontaneous or traumatic) necessitating treatment with bypass factor during the 6 months prior to Enrollment into Observational Phase and willing to continue to receive on-demand treatment during the Observational Phase.
* Participants who have documented inhibitors while on factor-replacement therapy but who do not meet the quantitative inhibitor criteria described in the prior bullet at the time of Screening (eg, participant with a previously documented high-titer inhibitor (≥5 BU/mL) and whose condition precludes re-challenge with FVIII or FIX replacement) may be considered for eligibility on a case-by-case basis with prior agreement from the Pfizer Medical Monitor
* Participants who meet the bleeding criteria noted above and who are on routine prophylaxis (defined as treatment by IV injection of bypass factor to prevent bleeding) and have demonstrated at least 80% compliance with scheduled prophylaxis regimen during the 6 months prior to enrollment, may be considered for eligibility on a case-by-case basis with discussion and agreement from the Pfizer medical monitor.

Exclusion Criteria

* Previous or current treatment for and/or history of coronary artery diseases, venous or arterial thrombosis or ischemic disease
* Known planned surgical procedure during the planned study period.
* Known hemostatic defect other than hemophilia A or B.
* Abnormal renal or hepatic function
* Current unstable liver or biliary disease
* Abnormal hematologic parameters
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator,
* Current routine prophylaxis with bypassing agent or non-coagulation non-factor- replacement therapy, or any previous treatment with a gene therapy product for treatment of hemophilia (participants treated with prophylaxis using bypassing agents or who had prior treatment with non-factor products may be considered on a case-by-case basis).
* Regular, concomitant therapy with immunomodulatory drugs

  - Ongoing or planned use of immune tolerance induction during the Observational Phase or Active Treatment Phase, or prophylaxis with FVIII or FIX replacement at any time after initiation of treatment with study intervention during the Active Treatment Phase
* Previous exposure to PF 06741086 during participation in studies B7841002 and B7841003.
* Participation in other studies involving investigational drug(s) or investigational vaccines within 30 days (or as determined by local requirements) or 5 half-lives prior to study entry and/or during study participation.
* CD4 cell count ≤200/uL if human immunodeficiency virus (HIV)-positive
* Screening ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Individuals with hypersensitivity or an allergic reaction to hamster protein or other components of the study intervention.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 12 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 189 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Annualized bleeding rate (ABR) of treated bleeding events | Through Observational Phase (6months) and Active Treatment Phase (12 months) for total of approximately 18 months
  Derived for each subject for each treatment period by using the following formula: ABR = number of bleeds requiring treatments/ (days on treatment period / 365.25)
Incidence and severity of thrombotic events | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Incidence of anti drug antibody [ADA] against PF-06741086 | Throughout Active Treatment Phase (12 months)
Incidence of clinically significant persistent neutralizing antibody [NAb] against PF-06741086 | Throughout Active Treatment Phase (12 months)
Incidence and severity of injection site reaction | Throughout Active Treatment Phase (12 months)
Number of participants with clinically significant changes from baseline in physical exam | From Baseline through Observation and Active Treatment (approximately 18 months)
Incidence of clinically significant laboratory value abnormalities | From Screening through Observation and Active Treatment (approximately 18 months)
Incidence of severe hypersensitivity and anaphylactic reactions | From Screening through Observational and Active Treatment (approximately 18 months)
Incidence of adverse events and serious adverse events | From screening through Observation and Active treatment (approximately 18 months)
Number of participants with clinically significant changes from baseline in vital signs | From Baseline through Observation and Active Treatment (approximately 18 months)
Incidence and severity of thromboticangiopathy | Throughout Active Treatment Phase (12 months)
Incidence of intravascular coagulation/consumption coagulopathy | Throughout Active Treatment Phase (12 months)

SECONDARY OUTCOMES:
Incidence of joint bleeds | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Incidence of spontaneous bleeds | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Incidence of target joint bleeds | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Incidence of total bleeds (treated and untreated) | Through Observational and Active Treatment Phases (18 Months)
Change from baseline in the Hemophilia Joint Health Score (HJHS) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Change from baseline in (Haemophilia Adult Quality of Life Questionnaire (Haem-A-QoL) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Change from baseline in Haemophilia Quality of Life Questionnaire for Children (Haemo-QoL) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Change from baseline in Hemophilia Adult Activities List (HAL) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Change from baseline in Hemophilia Pediatric Activities List (PedHAL) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Patient Global Impression of Change - Hemophilia (PGIC-H) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months
Change from baseline in EuroQol 5 Dimensions 5 Level (EQ-5D-5L) | Through Observational Phase (6 months) and Active Treatment Phase (12 months) for total of approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (4):
  - USF Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Northwell Health HTC, New Hyde Park, New York
  - Washington Institute for Coagulation, Seattle, Washington
- Bulgaria (2):
  - National Specialized Hospital for the Active Treatment of Hematological Diseases - EAD, Sofia, Sofia
  - UMHAT "Prof.Dr. Stoyan Kirkovich", Stara Zagora
- Canada (4):
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - McMaster Children's Hospital, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
- China (5):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- Hôpital Necker Enfants Malades, Paris, France
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- India (4):
  - Nirmal Hospital Pvt, Ltd, Surat, Gujarat
  - Sahyadri Clinical Research and Development Center, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu
- Italy (3):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Milan
  - Università degli Studi di Perugia, Azienda Ospedaliera di Perugia, Ospedale Santa Maria della, Perugia, PERUGIA
  - Università degli Studi di Roma "Sapienza"-Policlinico Umberto I, Roma, RM
- Japan (4):
  - Nagoya University Hospital - Transfusion Medicine, Nagoya, Aichi-ken
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Saitama Medical University Hospital, Iruma-gun, Saitama
- Mexico (2):
  - Hospital Universitario "Dr Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro Multidisciplinario para el Desarrollo Especializado de la Inv. Clínica en Yucatán, S.C.P., Mérida, Yucatán
- Sultan Qaboos University Hospital, Muscat, Oman
- FGBOU VO "Samara State Medical University" of MoH of Russia, Samara, Russia
- Saudi Arabia (2):
  - King Abdulaziz University Hospital, Jeddah
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Institute for Mother and Child healthcare "Dr Vukan Cupic", Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa
- South Korea (3):
  - Kyungpook National University Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital At Gangdong, Seoul
- Spain (5):
  - Hospital Universitario A Coruna, A Coruña, A CORUNA
  - Hospital Universitario Vall d´Hebron, Barcelona, BARCELONA
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario de Salamanca, Salamanca, SALAMANCA
  - Hospital Universitario Miguel Servet, Zaragoza, ZARAGOZA
- Taiwan (2):
  - ChangHua Christian Hospital, Changhua, CHANGHUA COUNTY
  - Taichung Veterans General Hospital, Taichung
- Turkey (Türkiye) (11):
  - Acibadem Adana Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Health Research and Practice Center Gazi Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Gaziantep University Sahinbey Research and Training Hospital, Gaziantep
  - Istanbul University Oncology Institute, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dr. Behcet Uz Child Diseases Surgery Education and Research Hospital, Izmir
  - Erciyes University Medical Faculty, Kayseri
  - Ondokuz Mayıs University Medical Faculty, Samsun
  - Karadeniz Technical University Medical Faculty, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Matino D, Acharya S, Taylor CT, Sun P, Agathon D, Raje S, Gould T, Palladino A, Mahlangu J. Efficacy and Safety of Marstacimab Prophylaxis in Hemophilia A/B With Inhibitors: Results from the Phase 3 BASIS Trial. Blood. 2025 Dec 6:blood.2025031065. doi: 10.1182/blood.2025031065. Online ahead of print. PMID 41351884
- [Derived] Matino D, Palladino A, Taylor CT, Hwang E, Raje S, Nayak S, McDonald R, Acharya SS, Mahlangu J, Jimenez-Yuste V, Choraria N, Yang R, Li CK, Al-Khabori M, Wali Y, Morales Adrian J, Park YS, Zulfikar OB, Teeter J. Marstacimab prophylaxis in hemophilia A/B without inhibitors: results from the phase 3 BASIS trial. Blood. 2025 Oct 2;146(14):1654-1663. doi: 10.1182/blood.2024027468. PMID 40608864
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841005